CLINICAL TRIAL: NCT03936829
Title: Cyclophosphamide in the Treatment of Panniculitis Associated Acquired Lipodystrophy Syndrome With Type 1 Diabetes
Brief Title: Cyclophosphamide in the Treatment of Associated Acquired Lipodystrophy Syndrome With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-PAALS&T1D
Record Dates: First submitted 2019-04-25; First posted 2019-05-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Lipodystrophy Acquired; Type1diabetes
Keywords: panniculitis associated acquired generalised lipodystrophy; cyclophosphamide
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Drug:Cyclophosphamide Dosage form: intravenous infusion Dosage: 500 mg/m2 of BSA Frequency: every 4 weeks Duration: 24 weeks
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Admitted to the hospital every 4 weeks. Cyclophosphamide was intravenously instilled (500mg mg/m2 of BSA) after contraindications are excluded. ECG monitoring will be taken during the medication. A total of 6 treatments will be performed.
  Other Names: CYC

SUMMARY:
This study evaluates the change of insulin resistance and glucose metabolism of patients with panniculitis associated acquired lipodystrophy syndrome and type 1 diabetes with the treatment of cyclophosphamide.

DETAILED DESCRIPTION:
Patients with panniculitis associated acquired lipodystrophy syndrome and type 1 diabetes have difficulty in blood glucose management due to the presence of both severe insulin resistance and complete insulin deficiency. It is often necessary to use insulin doses several times that of other children of the same age with type 1 diabetes.

Since autoimmune response is the main cause of panniculitis associated acquired lipodystrophy syndrome, immunosuppressive agents can suppress immune response, prevent and alleviate the progression of panniculitis and acquired lipodystrophy syndrome, and improve insulin resistance caused by subcutaneous fat deficiency.

Cyclophosphamide is a classic immunosuppressive agent. This study hopes to improve insulin resistance of patients with panniculitis associated acquired lipodystrophy syndrome and type 1 diabetes by cyclophosphamide treatment, thereby reducing insulin dosage and improving glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of type 1 diabetes mellitus: clinical manifestations of typical diabetes mellitus include polyphagia, polyuria, weight loss, or diabetic ketoacidosis, confirmed by blood sugar level, islet function and autoimmune antibody.
2. Meet the diagnostic criteria for panniculitis: fat biopsy suggests inflammatory infiltration.
3. Meet the diagnostic criteria for acquired lipodystrophy syndrome: childhood onset, clinically no nutritional deficiency or catabolism, systemic or partial subcutaneous fat reduction, genetic testing to exclude congenital lipodystrophy syndrome; low leptin level and autoantibodies can aid in diagnosis.

Exclusion Criteria:

1. Mature and effective treatment methods are available.
2. HIV, HBV and HCV were positive.
3. A the active period of infection.
4. At the active stage of malignant tumors.
5. Combination of other fatal diseases.
6. Existence of mental and psychological diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Average daily insulin dosage | week 21
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the last cyclophosphamide treatment, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)

SECONDARY OUTCOMES:
Average daily insulin dosage | week 1
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the first cyclophosphamidethe, blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | week 5
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the 2nd cyclophosphamide, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | week 9
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the 3rd cyclophosphamide, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | week 13
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the 4th cyclophosphamide, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | week 17
  Average daily insulin dosage of continuous three days (the average of the 1st, 2nd and 3rd days' insulin requirements after the 5th cyclophosphamide, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | from the completion of treatment to 3 months
  Average daily insulin dosage of continuous three days (the average of 3 days' insulin requirements 3 months after the last cyclophosphamide treatment, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | from the completion of treatment to 6 months
  Average daily insulin dosage of continuous three days (the average of 3 days' insulin requirements 6 months after the last cyclophosphamide treatment, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | from the completion of treatment to 9 months
  Average daily insulin dosage of continuous three days (the average of 3 days' insulin requirements 9 months after the last cyclophosphamide treatment, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
Average daily insulin dosage | from the completion of treatment to 12 months
  Average daily insulin dosage of continuous three days (the average of 3 days' insulin requirements 12 months after the last cyclophosphamide treatment, the blood glucose meets the ISPAD guideline as premeal 4.0-7.0 mmol/L, postmeal 5.0-10.0 mmol/L, prebed 4.4-7.8 mmol/L)
HbA1c level | week 1
  HbA1c level
HbA1c level | week 5
  HbA1c level
HbA1c level | week 9
  HbA1c level
HbA1c level | week 13
  HbA1c level
HbA1c level | week 17
  HbA1c level
HbA1c level | week 21
  HbA1c level
HbA1c level | from the completion of treatment to 3 months
  HbA1c level
HbA1c level | from the completion of treatment to 6 months
  HbA1c level
HbA1c level | from the completion of treatment to 9 months
  HbA1c level
HbA1c level | from the completion of treatment to 12 months
  HbA1c level

CONTACTS AND LOCATIONS:
Overall Officials: Feihong Luo, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebastchi J, Ajluni N, Neidert A, Oral EA. A Report of Three Cases With Acquired Generalized Lipodystrophy With Distinct Autoimmune Conditions Treated With Metreleptin. J Clin Endocrinol Metab. 2015 Nov;100(11):3967-70. doi: 10.1210/jc.2015-2589. Epub 2015 Sep 21. PMID 26390101
- [Background] Kumar R, Pilania RK, Bhatia A, Dayal D. Acquired generalised lipodystrophy and type 1 diabetes mellitus in a child: a rare and implacable association. BMJ Case Rep. 2018 Aug 3;2018:bcr2018225553. doi: 10.1136/bcr-2018-225553. PMID 30076164
- [Background] Gupta N, Asi N, Farah W, Almasri J, Barrionuevo P, Alsawas M, Wang Z, Haymond MW, Brown RJ, Murad MH. Clinical Features and Management of Non-HIV-Related Lipodystrophy in Children: A Systematic Review. J Clin Endocrinol Metab. 2017 Feb 1;102(2):363-374. doi: 10.1210/jc.2016-2271. PMID 27967300
- [Background] Carroll M, Mellick N, Wagner G. Dermatomyositis panniculitis: a case report. Australas J Dermatol. 2015 Aug;56(3):224-6. doi: 10.1111/ajd.12172. Epub 2014 Apr 1. PMID 24689899
- [Background] Li S, Yang H, Guo P, Ao X, Wan J, Li Q, Tan L. Efficacy and safety of immunosuppressive medications for steroid-resistant nephrotic syndrome in children: a systematic review and network meta-analysis. Oncotarget. 2017 Aug 21;8(42):73050-73062. doi: 10.18632/oncotarget.20377. eCollection 2017 Sep 22. PMID 29069848
- [Background] Brown RJ, Meehan CA, Cochran E, Rother KI, Kleiner DE, Walter M, Gorden P. Effects of Metreleptin in Pediatric Patients With Lipodystrophy. J Clin Endocrinol Metab. 2017 May 1;102(5):1511-1519. doi: 10.1210/jc.2016-3628. PMID 28324110
- [Background] Chong AY, Lupsa BC, Cochran EK, Gorden P. Efficacy of leptin therapy in the different forms of human lipodystrophy. Diabetologia. 2010 Jan;53(1):27-35. doi: 10.1007/s00125-009-1502-9. Epub 2009 Sep 2. PMID 19727665
- [Background] Joffe BI, Panz VR, Raal FJ. From lipodystrophy syndromes to diabetes mellitus. Lancet. 2001 May 5;357(9266):1379-81. doi: 10.1016/S0140-6736(00)04616-X. No abstract available. PMID 11356429
- [Background] Hussain I, Patni N, Garg A. Lipodystrophies, dyslipidaemias and atherosclerotic cardiovascular disease. Pathology. 2019 Feb;51(2):202-212. doi: 10.1016/j.pathol.2018.11.004. Epub 2018 Dec 27. PMID 30595509
- [Background] Weingartner JS, Zedek DC, Burkhart CN, Morrell DS. Lupus erythematosus panniculitis in children: report of three cases and review of previously reported cases. Pediatr Dermatol. 2012 Mar-Apr;29(2):169-76. doi: 10.1111/j.1525-1470.2011.01544.x. Epub 2011 Nov 8. PMID 22066977
- [Background] Diker-Cohen T, Cochran E, Gorden P, Brown RJ. Partial and generalized lipodystrophy: comparison of baseline characteristics and response to metreleptin. J Clin Endocrinol Metab. 2015 May;100(5):1802-10. doi: 10.1210/jc.2014-4491. Epub 2015 Mar 3. PMID 25734254
- [Background] Ale'ed A, Alsonbul A, Al-Mayouf SM. Safety and efficacy of combined cyclophosphamide and rituximab treatment in recalcitrant childhood lupus. Rheumatol Int. 2014 Apr;34(4):529-33. doi: 10.1007/s00296-013-2896-8. Epub 2013 Nov 12. PMID 24218286
- [Background] Park JY, Chong AY, Cochran EK, Kleiner DE, Haller MJ, Schatz DA, Gorden P. Type 1 diabetes associated with acquired generalized lipodystrophy and insulin resistance: the effect of long-term leptin therapy. J Clin Endocrinol Metab. 2008 Jan;93(1):26-31. doi: 10.1210/jc.2007-1856. Epub 2007 Oct 16. PMID 17940115

DOCUMENTS (3):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03936829/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03936829/SAP_001.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03936829/ICF_002.pdf